CLINICAL TRIAL: NCT07206953
Title: Effects of the Peer Functional Relationship Enhancement Program on Early Adolescents' Bullying Attitudes, Peer Relationships, Self-Efficacy, and Critical Thinking Skills
Brief Title: Peer Relationship Program: Effects on Bullying, Peer Relations, Self-Efficacy, and Critical Thinking
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hilal Mercan Akcay (Other)
Responsible Party: Sponsor-Investigator, Hilal Mercan Akcay, Lecturer in Child Development (Medipol University), Medipol University
Organization: Medipol University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E-68552689-302.08-00003617500
Record Dates: First submitted 2025-09-24; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Bullying
Keywords: Peer Relationships; Bullying Prevention; Early Adolescents; Group Intervention; Self-Efficacy; Critical Thinking; Psychoeducational Program
MeSH Terms: conditions — Bullying

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either an intervention group, which receives the Peer Relationship Enhancement Program, or a control group, which receives no intervention. Both groups are followed concurrently to compare outcomes.
Masking Description: Not applicable; this is an open-label study with no masked parties.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: Peer Relationship Enhancement Program (Experimental): Participants in this group receive the Peer Relationship Enhancement Program, consisting of nine weekly sessions focused on cooperative activities, role-play, and creative exercises designed to strengthen peer relationships, improve bullying attitudes, self-efficacy, and critical thinking skills.
  Interventions: Behavioral: Peer Functional Relationship Enhancement Program
- Control Group: No Intervention (No Intervention): Participants in this group do not receive any intervention and continue with their usual school activities. They serve as a comparison to evaluate the effects of the program.

INTERVENTIONS:
Behavioral: Peer Functional Relationship Enhancement Program — The Peer Functional Relationship Enhancement Program is a 9-week psychoeducational intervention for early adolescents. It consists of weekly group sessions that include cooperative activities, role-play, and creative exercises designed to strengthen peer relationships, improve attitudes toward bullying, enhance self-efficacy, and develop critical thinking skills. This program is structured and standardized to ensure consistent delivery across participants and is distinct from other behavioral or social skills programs targeting similar age groups.
  Arms: Intervention Group: Peer Relationship Enhancement Program

SUMMARY:
This study examines the effects of a Peer Relationship Enhancement Program on early adolescents' attitudes toward bullying, friendships, self-efficacy, and critical thinking skills. Participants will be early adolescents aged 11-12 years attending secondary schools. The program consists of 9 weekly group sessions with activities aimed at strengthening peer relationships and social skills. Assessments will be conducted before and after the program. The study is expected to help improve participants' self-efficacy, friendships, and taking an effective stance against bullying, critical thinking abilities.

DETAILED DESCRIPTION:
In Turkey, correlational research has been conducted over the last five years, with almost no experimental studies. Correlational studies have been conducted primarily with kindergarten and high school groups. Research indicates that there is no preventive research aimed at strengthening peer relationships among pre-adolescent children in middle school regarding their attitudes toward peer bullying. Consequently, these studies, both international and domestic, demonstrate that functional peer relationships, attitudes toward bullying, self-efficacy, and critical thinking skills are not addressed together. Therefore, the planned study is highly original and will contribute to existing scientific knowledge. Because peer bullying is an environmental risk factor that significantly impacts peer relationships, seven secondary schools affiliated with the Ministry of National Education in the Sapanca district of Sakarya province constitute the population of the study. This study, which will examine the effects of the Strengthening Functional Peer Relationships Program developed for pre-adolescent children on children's attitudes toward bullying, peer relationships, self-efficacy levels, and critical thinking skills, will utilize a pre-test, post-test, control group experimental design that requires measurements in control and experimental groups before and after the training. The study sample consisted of 48 6th-grade middle school students (ages 11-12) aged 11-12 who agreed to participate in the study. Before developing the Strengthening Functional Peer Relationships Program for pre-adolescent children, a needs assessment was conducted to identify topics in which they needed support regarding peer relationships, based on teachers' observations, to ensure the program was appropriate for the children's needs. Module topics were then determined, and an "Expert Opinion Form" prepared by the researcher to evaluate the outcomes and indicators was sent to five experts working in the field and finalized based on their opinions. The 9-week module content was developed in line with the outcomes and indicators. The final version was developed by consulting seven experts in the field. Modules last a minimum of 40 and a maximum of 90 minutes. Throughout the implementation of the training program, students were actively involved in the process using games, collaborative group work, question-and-answer, drawing, pantomime, brainstorming, storytelling, drama, observation, role-playing, reflective writing, mind mapping, scamper technique, problem-based learning, station technique, visually supported presentation, case study analysis, scenario-based group work, visual production, interactive storytelling, and art-based creative expression methods. SPSS will be used to analyze the research data. After examining outliers, the Shapiro-Wilk test will be applied to test for normal distribution. If the data are normally distributed, the independent samples t-test will be performed for paired groups, and the Anova test will be performed for groups of three or more. If the data are not normally distributed, the Mann-Whitney U test will be performed for paired groups, and the Kruskal-Willis H test will be performed for groups of three or more. It is thought that the thesis study will meet the need of the Ministry of National Education to prevent peer bullying in secondary schools.

ELIGIBILITY:
Inclusion Criteria:

* Early adolescents aged 11-12 years and currently in 6th grade
* No medical diagnosis or condition that would prevent participation
* Voluntary participation of the child in the study
* Parental/guardian consent obtained
* Ability to attend sessions regularly throughout the program

Exclusion Criteria:

* Any diagnosed cognitive or developmental disorder that would prevent participation in group activities
* Previous participation in a similar peer relationship program
* Lack of parental/guardian consent

Ages: 11 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-11-03 (Estimated); Study Completion 2025-12-08 (Estimated)

PRIMARY OUTCOMES:
Bullying Attitudes | Pre- and post-intervention (9 weeks)
  Changes in attitudes towards bullying among young people in early adolescence will be measured with the validated Attitudes Towards Bullying Scale.15-item, 3-point Likert scale: 1 = Agree, 2 = Neutral, 3 = Disagree. Total score range: 15-45 points (higher scores indicate more positive attitudes toward peers). Subscales: Approving Attitude (4 items, items 1-4): 4-12 points. Rejecting Attitude (5 items, items 5-9, reverse scored): 5-15 points. Neutral Attitude (6 items, items 10-15): 6-15 points.

SECONDARY OUTCOMES:
Peer Relationships | Pre- and post-intervention (9 weeks)
  Changes in peer relationships of young people in early adolescence will be measured with the validated Peer Relationship Scale for Children and Adolescents.29-item, 5-point Likert scale: 1 = Strongly Disagree, 2 = Disagree, 3 = Neutral, 4 = Agree, 5 = Strongly Agree. Total score range: 29-145 points (higher scores indicate better peer relationships). Subscales: Closeness (13 items: 1-13): 13-65 points. Popularity (4 items: 14-17): 4-20 points. Trust (7 items: 18-24): 7-35 points. Understanding (5 items: 25-29): 5-25 points.
Self-Efficacy | Pre- and post-intervention (9 weeks)
  Changes in self-efficacy of young people in early adolescence will be measured with the validated Self-Efficacy for Alternative Behaviors Towards Aggression Scale. 7-item, 5-point Likert scale:
  1 = Strongly Agree, 2 = Generally Agree, 3 = Sometimes Agree, 4 = Rarely Agree, 5 = Never Agree. All items are reverse scored, so higher scores indicate higher self-efficacy. Total score range: 7-35 points. Single-dimension scale (unidimensional).
Critical Thinking Skills | Pre- and post-intervention (9 weeks)
  Changes in critical thinking skills of young people in early adolescence will be measured with the validated Critical Thinking Disposition Scale for Middle School Students. 21-item, 5-point Likert scale: 1 = Never, 2 = Rarely, 3 = Sometimes, 4 = Often, 5 = Always. Total score range: 21-105 points (higher scores indicate higher critical thinking skills). Subscales: Dialectical Thinking (12 items: 1,2,3,5,6,7,8,9,12,14,16,17): 12-60 points. Disposition (4 items: 18,19,20,21): 4-20 points. Analysis (5 items: 4,10,11,13,15): 5-25 points

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Mercan Akçay, PhD Cand., Principal Investigator — Medipol University
Locations (1):
- Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No